CLINICAL TRIAL: NCT02745145
Title: A Phase II, Randomized, Double-blind, Placebo Controlled, Parallel-group, Multicenter Trial to Evaluate the Efficacy and Safety of Abituzumab in Subjects With Systemic Sclerosis-associated Interstitial Lung Disease (SSc-ILD)
Brief Title: Abituzumab in SSc-ILD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulties experienced in identifying participants who meet the eligibility criteria of the trial.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMR 200017-014; 2015-005023-11 (EudraCT Number)
Record Dates: First submitted 2016-04-15; First posted 2016-04-20 (Estimated); Results first posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-05

CONDITIONS: Systemic Sclerosis-associated Interstitial Lung Disease
Keywords: Double-Blind Method; Interstitial Lung Diseases; Systemic Scleroderma; Abituzumab; Mycophenolate; Efficacy, Safety
MeSH Terms: conditions — Lung Diseases, Interstitial; Scleroderma, Systemic | interventions — Abituzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Abituzumab 1500 milligram (mg) (Experimental)
  Interventions: Drug: Abituzumab 1500 mg
- Abituzumab 500 mg (Experimental)
  Interventions: Drug: Abituzumab 500 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abituzumab 1500 mg — Participants received Abituzumab 1500 mg administered as an intravenous infusion for 1 hour every 4 weeks up to Week 64.
  Arms: Abituzumab 1500 milligram (mg)
Drug: Abituzumab 500 mg — Participants received Abituzumab 500 mg administered as an intravenous infusion for 1 hour every 4 weeks up to Week 64.
  Arms: Abituzumab 500 mg
Drug: Placebo — Participants received Placebo matched to Abituzumab administered as an intravenous infusion for 1 hour every 4 weeks up to Week 64.
  Arms: Placebo

SUMMARY:
The purpose of this trial was to compare two doses of abituzumab with placebo and determine whether abituzumab was more effective, safer, would be better tolerated and could provoke better immune response than placebo in the treatment of participants with SSc-ILD who already receive constant doses of mycophenolate.

ELIGIBILITY:
Inclusion Criteria:

* Participants were eligible for this trial if they fulfill all of the following inclusion criteria:
* Female or male participants aged between 18 and 75 years of age who provide informed written consent.
* Participants fulfilling the 2013 American College of Rheumatology (ACR) /European League Against Rheumatism criteria for classification of systemic sclerosis (SSc).
* Disease duration of less than (<) 7 years from first non-Raynaud's symptom.
* Participants who had been taking the same mycophenolate regimen (stable dose) in a range of 1.5 to 3 gram (g)/day of Mycophenolate mofetil (MMF) or 1080 to 2160 milligram/day (mg/day) of MPS for at least 2 months prior to the Screening Visit and continued through Day 1 of the Treatment Period, of the lung on HRCT according to central reading.
* According to central readings: Diffusion capacity of the lung for carbon monoxide (DLCO) greater than or equal to (>=) 30 percent (%) predicted, Forced vital capacity (FVC) 40% to 85% predicted, and a ratio of FVC % predicted to DLCO % predicted >=1.8 is acceptable if right heart catheterization within 3 months of screening revealed no pulmonary hypertension. If these criteria were met, then High-resolution computed tomography (HRCT) of lungs will be performed, and must show at least 5% fibrosis for participants to be eligible.
* Female participants of childbearing potential must use a highly effective method of contraception to prevent pregnancy for 4 weeks before randomization and must agree to continue to practice adequate contraception for the duration of their participation in the trial (up to the last Safety Follow-Up Visit). For the purposes of this trial, women of childbearing potential were defined as "All female participants after puberty unless they were post-menopausal for at least 2 years or weresurgically sterile." Highly effective contraception is defined as 2 barrier methods (eg, female diaphragm and male condoms); or 1 barrier method with at least one of the following: spermicide, a hormonal method, or an intrauterine device. Note that because mycophenolate affects the metabolism of oral contraceptives and may reduce their effectiveness, women receiving mycophenolate who were using oral contraceptives for birth control should employ an additional contraceptive method (for example, male or female barrier method).

Exclusion Criteria:

* Any condition that in the Investigator's opinion constitutes an inappropriate risk or a contraindication for participation in the trial or that could interfere with the trial objectives, conduct, or evaluation.
* Renal impairment (glomerular filtration rate [GFR] <45 mL/minute (min)/1.73 square meter (m^2) as calculated by the Modification of Diet in Renal Disease equation) calculated as follows: GFR (mL/min per 1.73 m^2) = 175*(standardized serum creatinine)^-1.154 * (age)^-0.203 * 1.212 (if black) * 0.742 (if female)
* Urine dipstick with >=3 plus protein and urine protein:creatinine ratio more than (>)2 mg/mg.
* Known diagnosis of obstructive lung disease/emphysema (Forced Expiratory Volume [FEV1]/FVC ratio <0.65) and/or significant emphysematous change on screening HRCT.
* Other clinically significant abnormalities on HRCT not attributable to scleroderma or emphysema as defined above.
* Known diagnosis of other significant respiratory disorders.
* Pulmonary hypertension that fulfills at least one of the following:

  * Current/planned treatment with systemic therapy targeted to Pulmonary arterial hypertension (PAH) or pulmonary hypertension;
  * History of transthoracic echocardiography showing at least one of the following: tricuspid regurgitation jet >2.8 m/sec, right atrial enlargement (major dimension >53 mm), right ventricular enlargement (mid cavity dimension >35 mm), moderate to severe left ventricular dysfunction;
  * N-terminal prohormone brain natriuretic peptide >3*Upper limit of normal (ULN)
  * Considered by the investigator to require initiation of systemic targeted PAH therapy.
* Current clinical diagnosis of another inflammatory connective tissue disease (eg, systemic lupus erythematosus, rheumatoid arthritis, ankylosing spondylitis, or dermato/polymyositis). Concomitant scleroderma-associated myopathy, fibromyalgia, and secondary Sjögren's were allowed.
* Suspected/confirmed significant aspiration within the previous 6 months, for example.

  * viral/bacterial/fungal infection
  * infection requiring hospitalization
  * Treatment with parenteral anti-infectives within 4 weeks prior/during Screening Period
  * Completion of oral anti-infectives within 2 weeks of Screening
  * Use of oral anti-infectives during Screening Period
  * Vaginal candidiasis
  * onychomycosis
  * chronically suppressed oral herpes simplex virus
  * Prophylaxis for Pneumocystis jiroveci pneumonia
* History of/positive Human immunodeficiency virus, hepatitis C antibody and/or polymerase chain reaction or Hepatitis B surface antigen and/or hepatitis B core antibody (total and/or Immunoglobulin M) antibody at screening.
* History of/current diagnosis of active tuberculosis (TB), or untreated latent TB infection (LTBI).
* Presence of uncontrolled or New York Heart Association Class 3 or 4 congestive heart failure.
* History of cancer, except adequately treated (ie, no evidence of recurrence within 5 years prior screening) basal cell/squamous cell carcinomas of the skin (≤3 total in lifetime) or carcinoma in situ of the cervix.
* Known hypersensitivity to abituzumab DS or DP.
* Current smoker (incl. e-cigarettes) / smoking within 4 weeks of screening.
* Use of agents other than mycophenolate considered by the Investigator to have immunomodulating, immunosuppressive, or potential scleroderma disease-modifying properties within 2 months of screening visit is not allowed (or 5 months prior to the Screening Visit for cyclophosphamide). Hydroxychloroquine or chloroquine were permitted if dose has been stable for at least 4 weeks before the screening visit.
* Use of systemic corticosteroids above 10 mg/day prednisone equivalent within 4 weeks prior until last dose of study drug. Inhaled and topical corticosteroids were permitted.
* Use of any biologic agent within 12 weeks or 5 half-lives, whichever is longer, of screening.
* History of anti-CD20 B-cell depleting therapy, eg, rituximab or ocrelizumab within 6 months prior to screening visit.
* Use of anticoagulant or antiplatelet agent (aspirin =<350 mg daily is permitted).
* Clinically significant or predefined abnormalities in lab tests:

  * Aspartate aminotransferase, Alanine aminotransferase or alkaline phosphatase level >2.5*ULN;
  * Total bilirubin >1.5*ULN (other than that due to known Gilbert's disease);
  * Hemoglobin <5.0 mmol/L (9 g/dL), white blood cell count <2.5*10^9/L, or platelets <100*10^9/L);
  * International normalized ratio or partial thromboplastin time >2.0*ULN;
  * Thyroid-stimulating hormone <0.01 or >=7.1 milli international units per litre (mIU/L).
* Inability to receive IV infusions.
* History of alcohol/drug abuse for 1 year prior screening.
* Pregnancy/breastfeeding/lactation within 3 months prior screening.
* History of thrombotic, thromboembolic, or abnormal bleeding events including concomitant antiphospholipid antibody syndrome. Participants with known lupus anticoagulant and/or anticardiolipin and/or anti-b2 glycoprotein antibodies alone should not be excluded.
* Legal incapacity/limited legal capacity.
* Receipt/planned live/attenuated vaccination within 12 weeks prior screening until 3 months after last dose of study drug. Seasonal influenza vaccination with inactivated vaccine formulation is permitted.
* Major surgery requiring hospitalization within 4 weeks prior screening, planned major surgery for the duration of the trial. Participants with lung resection.
* History of/planned major organ or hematopoietic stem cell/marrow transplant.
* Severe gastrointestinal disease requiring parenteral nutrition. Other protocol defined exclusion criteria could apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., a business of Merck KGaA, Darmstadt, Germany
Locations (55):
- United States (18):
  - Research site 1, Los Angeles, California
  - Research site, Los Angeles, California
  - Research site, Farmington, Connecticut
  - Research site, Washington D.C., District of Columbia
  - Research site, Orlando, Florida
  - Research site, Weston, Florida
  - Research site, Chicago, Illinois
  - Research site 1, Boston, Massachusetts
  - Research site 2, Boston, Massachusetts
  - Research site, Ann Arbor, Michigan
  - Research site, New Brunswick, New Jersey
  - Research site, Great Neck, New York
  - Research site 1, New York, New York
  - Research site 2, New York, New York
  - Research site, Portland, Oregon
  - Research site, Nashville, Tennessee
  - Research site, Dallas, Texas
  - Research site, Houston, Texas
- Argentina (6):
  - Research site 1, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Research site 2, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Research site 3, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Research site, San Fernando, Buenos Aires
  - Research site, San Miguel de Tucumán, Tucumán Province
  - Research site, San Juan
- Australia (2):
  - Research site, Camperdown, New South Wales
  - Research site, Woodville South, South Australia
- Canada (2):
  - Research site, Vancouver, British Columbia
  - Research site, Toronto, Ontario
- Israel (6):
  - Research site, Haifa
  - Research site, Jerusalem
  - Research site, Kfar Saba
  - Research site, Petah Tikva
  - Research site, Ramat Gan
  - Research site, Tel Aviv
- Italy (9):
  - Research site, Torrette, Ancona
  - Research site, Rozzano, Milano
  - Research site 1, Milan
  - Research site 2, Milan
  - Research site, Napoli
  - Research site, Pisa
  - Research site, Reggio Emilia
  - Research site 1, Roma
  - Research site 2, Roma
- Poland (4):
  - Research site, Gdansk
  - Research site, Lodz
  - Research site 1, Warsaw
  - Research site 2, Warsaw
- Spain (2):
  - Research site, Madrid
  - Research site, Valladolid
- United Kingdom (6):
  - Research site, Cambridge, Cambridgeshire
  - Research site, London, Greater London
  - Research site, Cannock, Staffordshire
  - Research site, Dundee, Tayside Region
  - Research site, Birmingham, West Midlands
  - Research site, Sheffield, West Midlands

REFERENCES:
- [Derived] Khanna D, Tashkin DP, Wells AU, Seibold JR, Wax S, Vazquez-Mateo C, Fleuranceau-Morel P, Damian D, Denton CP. STRATUS: A Phase II Study of Abituzumab in Patients With Systemic Sclerosis-associated Interstitial Lung Disease. J Rheumatol. 2021 Aug;48(8):1295-1298. doi: 10.3899/jrheum.191365. Epub 2020 Oct 1. PMID 33004536

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study enrolled 24 participants and was early terminated due to the difficulties experienced in identifying participants who meet the eligibility criteria of the trial.
Groups:
- Abituzumab 500 Milligrams (mg): Participants received Abituzumab 500 mg administered as an intravenous infusion for 1 hour every 4 weeks up to Week 64.
Period: Overall Study
Arm/Group | Placebo | Abituzumab 500 Milligrams (mg) | Abituzumab 1500 mg
Started | 10 | 5 | 9
Completed | 0 | 0 | 0
Not Completed | 10 | 5 | 9
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Progressive disease | 0 | 0 | 1
Not completed — Withdrew consent | 1 | 1 | 1
Not completed — Study Termination | 8 | 3 | 7

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAF) included all participants who received at least 1 dose of abituzumab (including placebo) and have at least 1 post dose safety assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Abituzumab 500 Milligrams (mg) | Abituzumab 1500 mg | Total
Number analyzed (Participants) | 10 | 5 | 9 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51 (10.6) | 60 (7.5) | 55 (7.8) | 55 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 7 | 19
  Male | 2 | 1 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 3 | 4
  Not Hispanic or Latino | 9 | 5 | 6 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 5 | 9 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Absolute Forced Vital Capacity (FVC) at Week 52
Description: FVC was the maximum amount of air exhaled from the lungs after taking the deepest breath possible. The FVC assessments were done using spirometry. Change from baseline in fvc at week 52 was reported.
Time Frame: Baseline, Week 52
Population: Modified intent-to-treat (mITT) population was defined as all randomized participants who received at least 1 dose of study drug (including placebo). Here, "Overall Number of Participants Analyzed" signified participants evaluable for the outcome measure. All participants for abituzumab 500 mg arm dropped out before the analysis was conducted.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Placebo | Abituzumab 500 mg | Abituzumab 1500 mg
Number analyzed (Participants) | 2 | 0 | 1
milliliters | -130 (56.6) |  | -50 (NA) — Standard deviation was not estimable as there was only one participant evaluable for the arm.

2. Secondary Outcome: Change From Baseline in Dyspnea as Measured by the Mahler's Transition Dyspnea Index (TDI) at Week 52
Description: Mahler's TDI was an interview-administered instrument that allows participants to assess their level of dyspnea which was assessed by functional impairment, magnitude of task and magnitude of effort. Scores for each subscale range from -3 to +3 so that the TDI focal score ranges from -9 (major deterioration) to +9 (major improvement). For all subscale scores and the TDI focal score a higher value indicates a better outcome.
Time Frame: Baseline, Week 52
Population: mITT population was defined as all randomized participants who receive at least 1 dose of study drug (including placebo). Here, "Overall Number of Participants Analyzed" signified number of participants evaluable for the outcome measure. All participants for abituzumab 500 mg arm dropped out before the analysis was conducted.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Abituzumab 500 mg | Abituzumab 1500 mg
Number analyzed (Participants) | 1 | 0 | 1
Score on a scale | 3 (NA) — Standard deviation was not estimable as there was only one participant evaluable for the arm. |  | 4 (NA) — Standard deviation was not estimable as there was only one participant evaluable for the arm.

3. Secondary Outcome: Absolute Change From Baseline in St. George Respiratory Questionnaire (SGRQ) Total Score at Week 52
Description: The SGRQ assesses health-related quality of life in participants with chronic pulmonary disease by evaluating 3 health domains: symptoms (distress caused by respiratory symptoms); activity (effects of disturbances on mobility and physical activity); and impacts (the effect of disease on factors such as employment, personal control of one's health, and need for medication). A composite total score is derived as the weighted sum of domain scores for symptoms, activity, and impact (0=the best possible score and 100=the worst possible score). A reduction in score of 4 units is generally recognized as a clinically meaningful improvement in quality of life.
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Abituzumab 500 mg | Abituzumab 1500 mg
Number analyzed (Participants) | 1 | 0 | 1
Scores on a scale | 6.4 (NA) — Standard deviation was not estimable as there was only one participant evaluable for the arm. |  | 1.4 (NA) — Standard deviation was not estimable as there was only one participant evaluable for the arm.

4. Secondary Outcome: Absolute Change From Baseline in Modified Rodnan Skin Score (mRSS) at Week 52 in Participants With Diffuse Cutaneous Skin Involvement at Baseline
Description: The Modified Rodnan Skin Score (mRSS) measures dermal skin thickness through the examination of 17 body areas: fingers, hands, forearms, arms, feet, legs, and thighs (in pairs), and face, chest, and abdomen. The skin score is evaluated by manual palpation in each of these areas. The skin score is 0 for uninvolved skin, 1 for mild thickening, 2 for moderate thickening, and 3 for severe thickening (hidebound skin). The total skin score is the sum of the skin scores of the individual areas where the minimum score is 0 and the maximum score is 51. A higher score indicates greater severity of disease.
Time Frame: Baseline, Week 52
Population: mITT diffuse cutaneous systemic sclerosis population from mITT analysis set who had diffuse cutaneous skin involvement at baseline. Here, "Overall Number of Participants Analyzed" signified participants evaluable for the outcome measure. All participants for abituzumab 500 mg and abituzumab 1500 mg arm dropped out before the analysis was conducted.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Abituzumab 500 mg | Abituzumab 1500 mg
Number analyzed (Participants) | 1 | 0 | 0
Scores on a scale | 0 (NA) — Standard deviation was not estimable as there was only one participant evaluable for the arm. |  |

5. Secondary Outcome: Absolute Change From Baseline in Quantitative Lung Fibrosis (QLF) in the Region of Highest Baseline Severity at Week 52
Description: Absolute change from baseline in QLF score at week 52 was calculated as the difference of the QLF score at week 52 minus the QLF score at baseline divided in the region of highest baseline severity at Week 52 .The QLF score itself ranges from 0 to 100, where greater values represent a greater amount of lung fibrosis and are considered a worse health status.
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Abituzumab 500 mg | Abituzumab 1500 mg
Number analyzed (Participants) | 2 | 0 | 1
Scores on a scale | 6.29 (2.638) |  | -2.27 (NA) — Standard deviation was not estimable as there was only one participant evaluable for the arm.

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time (in months) from randomization to death. Data has been presented in terms of number participants who died and number of censored participants.
Time Frame: Time from date of randomization until death, assessed up to 2 years
Population: mITT population was defined as all randomized participants who receive at least 1 dose of study drug (including placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Abituzumab 500 mg | Abituzumab 1500 mg
Number analyzed (Participants) | 10 | 5 | 9
Participants
  Number of deaths | 0 | 1 | 0
  Number for censored | 10 | 4 | 9

7. Secondary Outcome: Number of Participants With Clinically Meaningful Progression of Systemic Sclerosis (SSc) by Meeting Criterion 1 (Interstitial Lung Disease [ILD])
Description: Clinically Meaningful Progression SSc-ILD was defined as one of the following (in the absence of causative intercurrent illness) on at least 2 occasions within approximately 4 weeks (per Outcome Measures in Rheumatology criteria): Relative decrease from baseline in forced vital capacity (FVC) % predicted greater than or equal to (>=)10%; Relative decrease from baseline in FVC % predicted of >=5% to less than (<) 10% and relative decrease from baseline in Diffusion capacity of the lung for carbon monoxide % predicted >=15%.
Time Frame: upto Week 52
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Abituzumab 500 mg | Abituzumab 1500 mg
Number analyzed (Participants) | 10 | 5 | 9
Participants | 0 | 0 | 2

8. Secondary Outcome: Number of Participants With Clinically Meaningful Progression of Systemic Sclerosis (SSc) by Meeting Criterion 2 (SSc Progression Other Than ILD)
Description: Clinically Meaningful Progression SSc other than ILD was defined as new onset of one or more of the following: Scleroderma renal crisis; Left ventricular failure (defined as ejection fraction <=45%); Pulmonary arterial hypertension requiring treatment.
Time Frame: upto Week 52
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Abituzumab 500 mg | Abituzumab 1500 mg
Number analyzed (Participants) | 10 | 5 | 9
Participants | 0 | 1 | 1

9. Secondary Outcome: Number of Participants With Clinically Meaningful Progression
Description: Participants meeting one or both of the below criteria was considered as having clinically meaningful disease progression. Clinically Meaningful SSc-ILD defined as one of the following (in the absence of causative intercurrent illness) on at least 2 occasions within approximately 4 weeks (per Outcome Measures in Rheumatology criteria): Relative decrease from baseline in forced vital capacity (FVC) % predicted greater than or equal to (>=)10%; Relative decrease from baseline in FVC % predicted of >=5% to less than (<) 10% and relative decrease from baseline in Diffusion capacity of the lung for carbon monoxide % predicted >=15%. Clinically Meaningful SSc progression other than ILD defined as new onset of one or more of the following: Scleroderma renal crisis; Left ventricular failure (defined as ejection fraction <=45%); Pulmonary arterial hypertension requiring treatment.
Time Frame: upto Week 52
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Abituzumab 500 mg | Abituzumab 1500 mg
Number analyzed (Participants) | 10 | 5 | 9
Participants | 0 | 1 | 2

10. Secondary Outcome: Number of Participants With Absolute Decrease From Baseline of FVC Percentage (%) Predicted Greater Than or Equal to (>=) 10% on 2 or More Consecutive Occasions at Least 4 Weeks Apart
Description: FVC is the maximum amount of air exhaled from the lungs after taking the deepest breath possible. The FVC assessments were done using spirometry.
Time Frame: upto Week 52
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Abituzumab 500 mg | Abituzumab 1500 mg
Number analyzed (Participants) | 10 | 5 | 9
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to 2 years
Arm/Group | Placebo | Abituzumab 500 Milligrams (mg) | Abituzumab 1500 mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/5 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/5 | 2/9
Other Adverse Events (participants affected / at risk) | 9/10 | 4/5 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | Abituzumab 500 Milligrams (mg) (N=5) | Abituzumab 1500 mg (N=9)
Disease progression (General disorders) | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Small fibre neuropathy (Nervous system disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | Abituzumab 500 Milligrams (mg) (N=5) | Abituzumab 1500 mg (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Eye pain (Endocrine disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 2
Generalised oedema (General disorders) | 0 | 1 | 0
Impaired healing (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 2
Pyrexia (General disorders) | 1 | 0 | 0
Multiple allergies (Immune system disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 4 | 0 | 0
Gastrointestinal bacterial overgrowth (Infections and infestations) | 1 | 0 | 0
Influenza (Gastrointestinal disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2
Onychomycosis (Infections and infestations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 1 | 0
Platelet count increased (Investigations) | 0 | 1 | 0
Protein urine present (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hot flush (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The analysis of outcome measures at Week 104 wasn't conducted as the study was terminated due to the difficulties experienced in identifying participants who meet the eligibility criteria of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT02745145/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT02745145/SAP_001.pdf